CLINICAL TRIAL: NCT01286298
Title: The Clinical Application of Diode Laser in Gingival Enlargement Related to Orthodontics
Brief Title: Diode Laser in Gingival Enlargement Related to Orthodontics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr. Tony Ngan-fat TO/ Master student, Orthodontics, Faculty of Dentistry, the University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 10-396
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Gingival Overgrowth
Keywords: diode laser; gingival enlargement; gingival overgrowth; gingival hyperplasia; orthodontics
MeSH Terms: conditions — Gingival Overgrowth; Gingival Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser gingivectomy (Experimental)
  Interventions: Procedure: Laser gingivectomy

INTERVENTIONS:
Procedure: Laser gingivectomy — Gingivectomy by diode laser
  Other Names: Biolase
Procedure: Laser gingivectomy — Diode laser gingivectomy for gingival enlargement
  Other Names: Biolase

SUMMARY:
Gingival enlargement is one of the most common soft tissue problems associated with fixed orthodontic treatment. The presence of orthodontic appliances impedes oral hygiene measures and alters the oral microbial ecosystem to a more pathogenic oral biofilm. Subsequent accumulation of plaque can contribute to development of chronic periodontal inflammation and can progress to gingival enlargement. Gingival enlargement inhibits hygiene measures, slows down orthodontic tooth movement and cause aesthetic and functional problems. Management of gingival enlargement by non-surgical periodontal treatment is considered to be most important and effective. Optimal plaque control can be maintained by meticulous brushing, flossing and professional scaling. However, motivation of maintaining oral hygiene can be disappointing in some patients. In cases that the enlarged gingivae became fibrous, surgical treatment can be considered.

Traditionally, gingivectomy was performed using scalpel under local infiltration. Since the first laser designed for dental use was introduced in 1989. Laser technology has continuously developed over the years and there are now many different types of dental lasers using a variety of wavelengths, e.g. Diode, Er:YAG, CO2 and Er,Cr:YSGG lasers. In orthodontics, various intraoral soft tissues surgical procedures may be required frequently, e.g. gingivectomy, gingivoplasty, fraenectomy, exposure of unerupted/ impacted/ partially erupted teeth. The use of laser has becoming more popular because the advantages of laser therapy are good haemostasis, excellent visualization of the operating field, fewer intra- and post-operative complications, bactericidal effect, no suture required, less scars, and better pain control with effects of reduced use of local anaesthesia and analgesic. Diode laser unit has the merits of compact size and relatively low price. Gingivectomy by diode laser may become an effective adjunctive treatment in orthodontic practice.

The aim of this study was to evaluate the clinical effectiveness of diode laser in the management of gingival enlargement related to orthodontic treatment.

DETAILED DESCRIPTION:
The null hypothesis: diode laser gingivectomy is not effective in gingival enlargement related to orthodontic treatment.

Outcome measures:

Plaque Index Gingival Index Bleeding on Probing Probing Pocket Depth Gingival Overgrowth Index Pain score by VAS

Inclusion criteria:

1. between 10-40 year-olds (inclusive).
2. gingival enlargement on the labial side of anterior teeth.
3. fit and healthy.
4. non-smokers.

ELIGIBILITY:
Inclusion Criteria:

1. between 10-40 year-olds (inclusive).
2. gingival enlargement on the labial side of anterior teeth.
3. fit and healthy.
4. non-smokers.

Exclusion Criteria:

1. gingival enlargement resolved after non-surgical periodontal treatment.
2. patients who refuse diode laser gingivectomy operation.
3. smokers
4. patients who are taking medications that may cause drug-associated gingival enlargement, e.g. calcium channel blockers, anticonvulsants or immunosuppressants.
5. patients with lingual orthodontic appliance.
6. pregnant or lactating women.
7. patients who are not competent in giving consents.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Gingival Overgrowth Index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tony NF TO, BDS, PDipGDS, Principal Investigator — The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, China